CLINICAL TRIAL: NCT01370577
Title: The Predictors for Asthma Control by Stepwise Treatment During 6 Months in Korean Elderly
Acronym: Prelude
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RKR-XXX-2011/1
Record Dates: First submitted 2011-06-01; First posted 2011-06-10 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
Keywords: Predictors for asthma control; Asthma Exacerbation rate; Mean frequency of PFT; sputum assessments; refill adherence(%); prescription persistence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Total 300 subjects who was diagnosed with asthma

SUMMARY:
The Predictors for asthma control by stepwise treatment during 6 months in Korean elderly

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or more, articulate in Korean
* Patients diagnosed with asthma, at least 1 year in duration.

Exclusion Criteria:

* Patients being followed-up for asthma treatment less than 1 year before baseline
* Patients taking immune therapy
* Patients previously enrolled/randomized in the present clinical trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged over 60 years, articulate in Korean, and diagnosed with asthma at least 1 year in duration
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics related to asthma control in the elderly | 6 months
Asthma exacerbation rate of the elderly during guideline-based stepwise treatments | 6 months

SECONDARY OUTCOMES:
1. Proportion of controlled, partially controlled, and controlled patients among the elderly patients with asthma in Korea | 6 months
2. Baseline characteristics related to asthma specific QOL in the elderly patients with asthma | 6 months
Mean frequency of PFT, sputum assessments, refill adherence(%), prescription persistence in elderly asthma for the last 1 year before study enrollment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hye Won Koo, Study Director — AstraZeneca Korea
Locations (5):
- South Korea (5):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Busan, Gyeonsangnam-do
  - Research Site, Changwon, Gyeonsangnam-do